CLINICAL TRIAL: NCT02963558
Title: ASPIRE: A Study Promoting Critical Illness Recovery in the Elderly
Brief Title: A Study Promoting Critical Illness Recovery in the Elderly
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00039558; 5UL1TR001420-03 (NIH); 1R03AG060076 (NIH)
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-05

CONDITIONS: Acute Respiratory Distress Syndrome; Critical Illness; Critical Care
MeSH Terms: conditions — Respiratory Distress Syndrome; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive in-bed cycle ergometry within 48 hours of randomization if safety criteria are met. The intervention arm will receive early physical therapy (PT). This PT will be performed according to a protocol of additional ICU and hospital-administered rehabilitation strategies that have been previously developed. Patients will receive 30 minutes of PT at least 5 times per week while conscious. If unconscious, subjects will only receive passive range of motion (PROM) for 10 repetitions per body part daily. Once conscious, subjects will progress through PT with an emphasis on ambulation. Therapy for the intervention arm patients will continue while on the floor. Outpatient therapy will be provided at the discretion of the patient's treating physicians.
  Interventions: Device: cycle ergometry
- Usual Care (No Intervention): The control group will receive usual care physical therapy as ordered by the treating team both in the ICU and on the floor through hospital discharge. These subjects will also receive therapy as outpatients only as ordered by their regular physicians.

INTERVENTIONS:
Device: cycle ergometry — The cycler will provide 3 different possible modes of cycling-passive, active-assisted, and active. The subject will start with passive cycling and may progress to active-assisted and active cycling.
  Other Names: MOTOmed
  Arms: Intervention

SUMMARY:
This proposal will test the hypothesis that EARLY application of a novel early rehabilitation therapy in critically ill patients will improve functional outcomes, and change the functional trajectory of this population. A pilot study of early mobilization with a cycle ergometer will be performed and translate into humans the pre-clinical mechanisms that may mediate the effects of early mobility. A second phase of the study was added in September 2019, which will focus on clinical outcomes.

DETAILED DESCRIPTION:
Patients will be randomized to intervention or control groups. Patients will receive therapies according to their group assignment until hospital discharge or day 28, whichever comes first.

The intervention group will receive in-bed cycle ergometry within 48 hours of randomization if safety criteria are met. In-bed cycle ergometry has been shown to be safe and feasible in the critically ill and is approved for use in this population. Subjects enrolled in the intervention arm will be screened at least 5 days per week to evaluate if they meet pre-defined safety criteria based on other studies of early mobilization and cycling in the Intensive Care Unit (ICU). Patients will be positioned in the semi-recumbent position for cycling as per ICU guidelines. The cycler will provide 3 different possible modes of cycling-passive, active-assisted, and active. The investigators will start with passive cycling and the patient may progress to active-assisted and active cycling. The goal duration of cycling will be 30 minutes. Subjects will receive in-bed cycling at least 5 times per week for the duration of the ICU stay or until day 14, whichever comes first. During cycling and therapy sessions, the physical therapist will also complete a case report form noting vital signs, level of mobilization, and other safety measures.

In addition to cycling, the intervention arm will receive early physical therapy (PT). This physical therapy will be performed according to a protocol of additional ICU and hospital-administered rehabilitation strategies that were previously developed. Patients will receive 30 minutes of Physical Therapy (PT) at least 5 times per week when they are conscious. If unconscious, subjects will only receive passive range of motion (PROM) for 10 repetitions per body part daily. Once conscious, subjects will progress through the different levels of PT with an emphasis on ambulation.

Physical therapy for the intervention arm patients will continue while hospitalized through day 28. Outpatient therapy will be provided at the discretion of the patient's treating physicians.

The control group will receive usual care physical therapy as ordered by the treating team both in the ICU and on the floor through hospital discharge. These subjects will also receive therapy as outpatients only as ordered by their physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55 years old
* Admission to Wake Forest Baptist Medical Center Medical Intensive Care Unit
* Acute Hypoxic respiratory failure on mechanical ventilation for <48 hours with a P:F ratio of <300 (or equivalent S:F ratio)
* Previously Functional (over past 3 months, as reported by proxy):

Physical Function: Able to walk 4 m (with or without assistive device)

Exclusion Criteria:

* Neuromuscular Disease
* Cardiopulmonary Arrest with return of spontaneous circulation <6 hrs
* Palliative Goals of Care; witholding life-sustaining therapy
* Elevated Intracranial Pressure (>20 mm Hg)
* BMI>45; absolute weight >= 150 kg
* Inability to cycle (including absent limbs, body length <1.5m, body habitus not fitting the cycle, inflammatory arthritis, significant joint problems including inability to bend arms/legs; pelvic and/or LE fracture, LE bypass surgery)
* Pregnancy
* Unable to speak English
* Use of continuous neuromuscular blockade
* Temporary Pacemaker or Swan Ganz catheter or femoral ECMO catheter/IABP
* Rhabdomyolysis with most recent CK >5000
* Clinical diagnosis of dementia on medication
* Moribund
* Possible Exclusion: If the patient is on spine precautions, a discussion with the spine team will be necessary to determine eligibility for the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Clark Files, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Herridge MS, Chu LM, Matte A, Tomlinson G, Chan L, Thomas C, Friedrich JO, Mehta S, Lamontagne F, Levasseur M, Ferguson ND, Adhikari NK, Rudkowski JC, Meggison H, Skrobik Y, Flannery J, Bayley M, Batt J, Santos CD, Abbey SE, Tan A, Lo V, Mathur S, Parotto M, Morris D, Flockhart L, Fan E, Lee CM, Wilcox ME, Ayas N, Choong K, Fowler R, Scales DC, Sinuff T, Cuthbertson BH, Rose L, Robles P, Burns S, Cypel M, Singer L, Chaparro C, Chow CW, Keshavjee S, Brochard L, Hebert P, Slutsky AS, Marshall JC, Cook D, Cameron JI; RECOVER Program Investigators (Phase 1: towards RECOVER); Canadian Critical Care Trials Group. The RECOVER Program: Disability Risk Groups and 1-Year Outcome after 7 or More Days of Mechanical Ventilation. Am J Respir Crit Care Med. 2016 Oct 1;194(7):831-844. doi: 10.1164/rccm.201512-2343OC. PMID 26974173
- [Background] Ely EW, Wheeler AP, Thompson BT, Ancukiewicz M, Steinberg KP, Bernard GR. Recovery rate and prognosis in older persons who develop acute lung injury and the acute respiratory distress syndrome. Ann Intern Med. 2002 Jan 1;136(1):25-36. PMID 11777361
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Denehy L, Skinner EH, Edbrooke L, Haines K, Warrillow S, Hawthorne G, Gough K, Hoorn SV, Morris ME, Berney S. Exercise rehabilitation for patients with critical illness: a randomized controlled trial with 12 months of follow-up. Crit Care. 2013 Jul 24;17(4):R156. doi: 10.1186/cc12835. PMID 23883525
- [Background] Moss M, Nordon-Craft A, Malone D, Van Pelt D, Frankel SK, Warner ML, Kriekels W, McNulty M, Fairclough DL, Schenkman M. A Randomized Trial of an Intensive Physical Therapy Program for Patients with Acute Respiratory Failure. Am J Respir Crit Care Med. 2016 May 15;193(10):1101-10. doi: 10.1164/rccm.201505-1039OC. PMID 26651376
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Background] Files DC, Liu C, Pereyra A, Wang ZM, Aggarwal NR, D'Alessio FR, Garibaldi BT, Mock JR, Singer BD, Feng X, Yammani RR, Zhang T, Lee AL, Philpott S, Lussier S, Purcell L, Chou J, Seeds M, King LS, Morris PE, Delbono O. Therapeutic exercise attenuates neutrophilic lung injury and skeletal muscle wasting. Sci Transl Med. 2015 Mar 11;7(278):278ra32. doi: 10.1126/scitranslmed.3010283. PMID 25761888
- [Background] Walsh TS, Salisbury LG, Merriweather JL, Boyd JA, Griffith DM, Huby G, Kean S, Mackenzie SJ, Krishan A, Lewis SC, Murray GD, Forbes JF, Smith J, Rattray JE, Hull AM, Ramsay P; RECOVER Investigators. Increased Hospital-Based Physical Rehabilitation and Information Provision After Intensive Care Unit Discharge: The RECOVER Randomized Clinical Trial. JAMA Intern Med. 2015 Jun;175(6):901-10. doi: 10.1001/jamainternmed.2015.0822. PMID 25867659
- [Background] Files DC, Sanchez MA, Morris PE. A conceptual framework: the early and late phases of skeletal muscle dysfunction in the acute respiratory distress syndrome. Crit Care. 2015 Jul 2;19(1):266. doi: 10.1186/s13054-015-0979-5. PMID 26134116
- [Background] Bakhru RN, Wiebe DJ, McWilliams DJ, Spuhler VJ, Schweickert WD. An Environmental Scan for Early Mobilization Practices in U.S. ICUs. Crit Care Med. 2015 Nov;43(11):2360-9. doi: 10.1097/CCM.0000000000001262. PMID 26308435
- [Background] Jolley SE, Dale CR, Hough CL. Hospital-level factors associated with report of physical activity in patients on mechanical ventilation across Washington State. Ann Am Thorac Soc. 2015 Feb;12(2):209-15. doi: 10.1513/AnnalsATS.201410-480OC. PMID 25565021
- [Background] Jolley SE, Regan-Baggs J, Dickson RP, Hough CL. Medical intensive care unit clinician attitudes and perceived barriers towards early mobilization of critically ill patients: a cross-sectional survey study. BMC Anesthesiol. 2014 Oct 1;14:84. doi: 10.1186/1471-2253-14-84. eCollection 2014. PMID 25309124
- [Background] Camargo Pires-Neto R, Fogaca Kawaguchi YM, Sayuri Hirota A, Fu C, Tanaka C, Caruso P, Park M, Ribeiro Carvalho CR. Very early passive cycling exercise in mechanically ventilated critically ill patients: physiological and safety aspects--a case series. PLoS One. 2013 Sep 9;8(9):e74182. doi: 10.1371/journal.pone.0074182. eCollection 2013. PMID 24040200
- [Background] Kho ME, Martin RA, Toonstra AL, Zanni JM, Mantheiy EC, Nelliot A, Needham DM. Feasibility and safety of in-bed cycling for physical rehabilitation in the intensive care unit. J Crit Care. 2015 Dec;30(6):1419.e1-5. doi: 10.1016/j.jcrc.2015.07.025. Epub 2015 Jul 29. PMID 26318234
- [Background] Parry SM, Berney S, Warrillow S, El-Ansary D, Bryant AL, Hart N, Puthucheary Z, Koopman R, Denehy L. Functional electrical stimulation with cycling in the critically ill: a pilot case-matched control study. J Crit Care. 2014 Aug;29(4):695.e1-7. doi: 10.1016/j.jcrc.2014.03.017. Epub 2014 Mar 26. PMID 24768534
- [Background] Needham DM, Korupolu R, Zanni JM, Pradhan P, Colantuoni E, Palmer JB, Brower RG, Fan E. Early physical medicine and rehabilitation for patients with acute respiratory failure: a quality improvement project. Arch Phys Med Rehabil. 2010 Apr;91(4):536-42. doi: 10.1016/j.apmr.2010.01.002. PMID 20382284

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 14 | 10
Completed | 13 | 9
Not Completed | 1 | 1
Not completed — Withdrawn by investigator | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 64 [59 to 70] | 71 [64.5 to 72.5] | 68 [61.25 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in the Intervention Arm Who Are Able to Undergo a Cycling Session
Description: Feasibility will be assessed by quantifying the ability to apply the MOTOmed device for at least a 15-minute session within 48 hours of randomization and meeting safety criteria.
Time Frame: up to 48 hours after randomization
Population: This outcome only pertains to the interventional arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 0
Participants | 13 | 0

2. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: Based on timed measures of standing balance, walking speed, and ability to rise from a chair. Scores range from 0-12. A higher score denotes a better outcome.
Time Frame: Intensive Care Unit (ICU) discharge (through study completion, on average day 10)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
score on a scale | 3 [0 to 5] | 1 [0 to 2]

3. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: Based on timed measures of standing balance, walking speed, and ability to rise from a chair. Score ranges from 0 to 12. A higher score denotes a better outcome.
Time Frame: Hospital discharge (through study completion, on average day 10)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
score on a scale | 3 [0 to 6] | 4.25 [1 to 7]

4. Secondary Outcome: Handgrip Strength
Description: Assessed with a Jamar hand-held dynamometer.
Time Frame: ICU Discharge, Hospital discharge (through study completion, on average day 10)
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
kilograms
  ICU Discharge | 11.33 [0 to 18.6] | 11.33 [7 to 21.33]
  Hospital Discharge | 14.33 [0 to 20] | 8.67 [0 to 18.67]

5. Secondary Outcome: Mobility Assessment Tool-short Form (MAT-sf)
Description: A scoring system from 30 to 80 with 80 meaning higher physcial function
Time Frame: Day 0, ICU discharge, Hospital discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
score on a scale
  Day 0 | 55.4 [37.7 to 64.7] | 49.12 [46.0 to 62.3]
  ICU Discharge | 42.8 [36.4 to 48.1] | 54.0 [49.1 to 62.1]
  Hospital Discharge | 45.4 [40.9 to 46.9] | 47 [42.8 to 50.0]

6. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: screening instrument for mild cognitive dysfunction; range 0-30; lower score means more cognitive impairment
Time Frame: hospital discharge, month 3, month 6
Population: Not adminstered at month 3 and month 6; no data collected for those time frames
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
score on a scale
  Hospital discharge | 18.5 [16.75 to 22.0] | 19 [15.5 to 23.5]
  Month 3: number analyzed (Participants) | 0 | 0
  Month 6: number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Quad Strength
Description: Measurement of quadriceps strength while sitting.
Time Frame: ICU Discharge, Hospital discharge
Measure: Median (Inter-Quartile Range); unit: newtons
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
newtons
  ICU Discharge | 11.6 [0 to 18.9] | 12.37 [4.97 to 22.4]
  Hospital Discharge | 12.9 [0 to 20.03] | 13.1 [0 to 18.97]

8. Secondary Outcome: Short Form-36
Description: Assesses quality of life. Score for each part of the questionnaire ranges from 0 to 100. Data will be collected for the following parts: Physical functioning, Role Limited Due to Physical Health, Role Limited Due to Emotional Problems, Energy/Fatigue, Emotional Well-being, Social Functioning, Pain, General Health. For each of these a higher score means better function/less impariment in regards to each item.
Time Frame: hospital discharge
Population: Only completed at hospital discharge; data not collected at any other time frame
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
score on a scale
  Physical Functioning | 15 [0 to 45] | 20 [5 to 20]
  Role Limited Due to Physical Health | 0 [0 to 0] | 0 [0 to 0]
  Energy/Fatigue | 0 [0 to 0] | 33.33 [0 to 66.67]
  Emotional Well-Being | 24 [0 to 72] | 56 [20 to 76]
  Social Functioning | 0 [0 to 12.5] | 0 [0 to 37.5]
  Pain | 22.5 [0 to 55] | 55 [0 to 77.5]
  General Health | 25 [0 to 60] | 25 [20 to 40]

9. Secondary Outcome: Muscle Ultrasound--tibialis Anterior Depth
Description: The study team is measuring the percentage of the size of the cross-sectional area of the tibialis anterior. Day 0 for everyone is 100% (starting point). The study team is measuring the percentage of that starting point at other time points.
Time Frame: day 0, day 3, day 5, ICU discharge, Hospital Discharge
Measure: Median (Inter-Quartile Range); unit: percentage of starting amount
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
percentage of starting amount
  Day 0 | 100 [100 to 100] | 100 [100 to 100]
  Day 3 | 94 [91 to 103] | 102 [99 to 104]
  Day 5 | 98 [94 to 102] | 102 [92 to 102]
  ICU Discharge | 102 [91 to 110] | 99 [90 to 103]
  Hospital Discharge | 94 [93 to 110] | 101 [98 to 102]

10. Secondary Outcome: Muscle Ultrasound--echogenicity in the Tibialis Anterior
Description: Obtain preliminary data to estimate the treatment effect size. Echogenicity is a measure called the "grey scale measure". Scores range from 0-255. A higher score is brighter/more white on ultrasound. A lower score is darker. Think of this as exposure on a black and white picture.
Time Frame: day 0, day 3, day 5, ICU discharge, Hospital Discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
units on a scale
  Day 0 | 76.07 (24.50) | 74.94 (24.50)
  Day 3 | 74.98 (24.64) | 73.62 (24.63)
  Day 5 | 78.03 (26.20) | 74.78 (24.90)
  ICU Discharge | 75.89 (25.06) | 73.31 (24.62)
  Hospital Discharge | 75.22 (25.75) | 73.30 (22.62)

11. Secondary Outcome: Muscle Ultrasound--muscle Depth Quadriceps
Description: The study team is measuring the percentage of the size of the cross-sectional area of the quadriceps. Day 0 for everyone is 100% (starting point). The study team is measuring the percentage of that starting point at other time points.
Time Frame: day 0, day 3, day 5, ICU discharge, Hospital Discharge
Measure: Median (Inter-Quartile Range); unit: percent of starting amount
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
percent of starting amount
  Day 0 | 100 [100 to 100] | 100 [100 to 100]
  Day 3 | 90 [84 to 110] | 94 [83 to 113]
  Day 5 | 102 [81 to 109] | 76 [69 to 87]
  ICU Discharge | 88 [80 to 94] | 80 [69 to 87]
  Hospital Discharge | 97 [69 to 104] | 87 [85 to 99]

12. Secondary Outcome: Muscle Ultrasound--muscle Size CSA of Rectus Femoris Muscle
Description: The study team is measuring the percentage of the size of the cross-sectional area of the rectus femoris. Day 0 for everyone is 100% (starting point). The study team is measuring the percentage of that starting point at other time points.
Time Frame: day 0, day 3, day 5, ICU discharge, Hospital Discharge
Measure: Median (Inter-Quartile Range); unit: percent of starting amount
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
percent of starting amount
  Day 0 | 100 [100 to 100] | 100 [100 to 100]
  Day 3 | 95 [77 to 105] | 95 [76 to 119]
  Day 5 | 91 [72 to 113] | 85 [75 to 95]
  ICU Discharge | 79 [66 to 83] | 84 [77 to 88]
  Hospital Discharge | 83 [72 to 93] | 95 [90 to 103]

13. Secondary Outcome: Muscle Ultrasound--echogenicity in the Rectus Femoris Muscle
Description: as for outcome 10
Time Frame: day 0, day 3, day 5, ICU discharge, Hospital Discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 13 | 9
units on a scale
  Day 0 | 73.34 (23.45) | 70.41 (23.08)
  Day 3 | 74.34 (25.73) | 67.73 (27.17)
  Day 5 | 71.78 (24.38) | 69.01 (23.29)
  ICU Discharge | 72.06 (26.03) | 64.50 (24.05)
  Hospital Discharge | 68.27 (25.39) | 63.62 (23.79)

14. Other Pre Specified Outcome: Accelerometer Activity Monitoring Results
Description: Used to determine activity.
Time Frame: Up through two weeks after discharge
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Number of Hospital Readmissions
Time Frame: up to 6 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Number of Emergency Department Visits
Time Frame: up to 6 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Number of Ventilator Free Days
Time Frame: Up to 28 days from hospital admission or hospital discharge, whichever is first
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Translational Outcomes
Description: MuRF1, NFKB, myofiber size and type, etc
Time Frame: up to 6 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Hospital Length of Stay
Description: Number of days
Time Frame: Hospital discharge (through study completion, on average day 10)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Mortality
Description: total number affected
Time Frame: up through 6 months post-discharge
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Intensive Care Unit (ICU) Length of Stay
Description: Number of days
Time Frame: ICU discharge (through study completion, on average day 7)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: through hospital discharge (an average of 10 days)
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/13 | 2/9
Serious Adverse Events (participants affected / at risk) | 4/13 | 2/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=13) | Usual Care (N=9)
exacerbation of underlying condition resulting in death (General disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT02963558/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT02963558/ICF_001.pdf